CLINICAL TRIAL: NCT00655135
Title: Phase 2 Randomized, Placebo-Controlled, Double-Blind, Parallel Group Study to Determine the Safety, Pharmacokinetics, and Effectiveness of LDP-02 in Patients With Mildly to Moderately Active Crohn's Disease
Brief Title: Phase 2 Study of the Safety and Efficacy of LDP-02 in Mildly to Moderately Active Crohn's Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Medical Monitor, Millennium Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L299-016
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — LDP-02; vedolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Patients were assigned to arms in a 1:1:1 ratio. Patients in this arm received placebo administered intravenously to patients on Day 1 and Day 29.
  Interventions: Drug: Placebo
- 2 (Experimental): Patients were assigned to arms in a 1:1:1 ratio. Patients in this arm received 0.5 mg/kg of LDP-02 administered intravenously to patients on Day 1 and Day 29.
  Interventions: Drug: LDP-02
- 3 (Experimental): Patients were assigned to arms in a 1:1:1 ratio. Patients in this arm received 2 mg/kg of LDP-02 administered intravenously to patients on Day 1 and Day 29.
  Interventions: Drug: LDP-02

INTERVENTIONS:
Drug: LDP-02 — Each patient in arms 2 & 3 received a single IV dose of study drug at 0.5 or 2.0 mg/kg LDP-02 on Days 1 and 29.
  Other Names: MLN0002, MLN02
  Arms: 2; 3
Drug: Placebo — Each patients in arm 1 received a single IV dose of placebo on Days 1 and 29.
  Other Names: MLN0002, MLN02
  Arms: 1

SUMMARY:
The objectives of this study were to assess the safety and tolerability of LDP-02 in patients with active Crohn's disease who were not receiving corticosteroids or immunosuppressives, to assess the ability of LDP-02 to reduce Crohn's disease activity, and to obtain pharmacokinetic (PK) and pharmacodynamic(PD)information for LDP-02 in patients with active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80, nonhospitalized, male or nonpregnant, nonlactating females voluntarily able to give informed consent.
* Crohn's disease of at least 6 months' duration.
* Endoscopic and/or histopathological and/or radiological documentation consistent with Crohn's disease obtained preferably within 24 months of screening.
* Crohn's disease involving the colon and/or the ileum.
* CDAI score from 220 to 400 (inclusive) at the time of the Screening visit. The CDAI must have remained between 220 and 400 after the 1-week Screening period for the patient to be eligible.
* Patients may have been receiving oral or topical 5-ASA compounds provided the dosage had been stable for at least the 14-day period before the Screening visit. Patients were to be maintained on the 5-ASA compound at a constant dose at least through Day 57.

Exclusion Criteria:

* Patients with evidence of current GI infection (bacterial or parasitic) or significant infection within 45 days of the screening visit.
* Patients with a serious underlying disease other than Crohn's disease including presence or history of malignancy (except basal cell carcinoma) and histological evidence of dysplasia.
* Patients with significantly impaired liver or renal function. This includes those with established chronic liver disease including hepatitis B or C.
* Patients with the laboratory abnormalities
* Patients using ethanol or consuming illicit drugs which, in the investigator's opinion, may interfere with compliance with the study procedures.
* Patients with active psychiatric problems which, in the investigator's opinion, may interfere with compliance with the study procedures.
* Patients who have previously received or who are currently receiving treatment with a monoclonal antibody.
* Patients receiving any investigational therapy, excluded medications as defined in protocol, or any approved therapy in an investigational protocol within 30 days prior to screening.
* Patients unable to attend all the study visits or comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2000-02; Primary Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was the proportion of patients with a clinical response, defined as a reduction from baseline in the CDAI score of at least 70 points at Day 57 | Days 1-57

REFERENCES:
- [Derived] Feagan BG, Greenberg GR, Wild G, Fedorak RN, Pare P, McDonald JW, Cohen A, Bitton A, Baker J, Dube R, Landau SB, Vandervoort MK, Parikh A. Treatment of active Crohn's disease with MLN0002, a humanized antibody to the alpha4beta7 integrin. Clin Gastroenterol Hepatol. 2008 Dec;6(12):1370-7. doi: 10.1016/j.cgh.2008.06.007. Epub 2008 Oct 1. PMID 18829392